CLINICAL TRIAL: NCT05106998
Title: Pattern of Nailfold Capillaroscopy Changes in Systemic Lupus Erythematosus Patients and Its Correlation With Anti-Uridin1-ribonucleoprotein Antibodies and Disease Activity
Brief Title: NFC Changes in SLE Patients and Its Correlation With Anti-U1RNPAntibodies and Disease Activity
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amera Imam Abdel - Ghany Ahmed, Resident doctor at Physical medicine ,Rheumatology and Rehabilitation department, Assiut University
Other Study IDs: NFC in SLE , Anti-U1RNP Ab
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: System Lupus Erythematosus
Keywords: nailfold capillaroscopy; anti-U1RNP antibodies; Disease activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Microscopic Angioscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Device: Yes

INTERVENTIONS:
Device: nailfold capillaroscopy — Nailfold capillaroscopy (NFC) is a non-invasive easily repeatable technique and the best method for morphological analysis of nutritional capillaries in the nailfold area

SUMMARY:
1. Detection of different pattern of nail fold capillary changes in SLE patient.
2. Correlation of nail fold capillary changes in SLE patients and Anti-U1RNP antibodies.
3. Correlation of nail fold capillary changes with SLE disease activity.
4. Frequency of nail fold capillary changes in SLE patients

DETAILED DESCRIPTION:
Systemic lupus erythematosus is a complex, multi-organ autoimmune disease . The presence of autoantibodies and circulating immune complexes can cause vasculitis and damage the endothelial cells, leading to multiple organ dysfunctions .The clinical manifestations of SLE include muco cutaneous, musculoskeletal system, cardiac, neurological, renal, hematologic, and vascular system involvement . Nail fold capillaroscopy (NFC) is a non-invasive easily repeatable technique and the best method for morphological analysis of nutritional capillaries in the nail fold area . Nail fold capillary changes are very common in patients with SLE. the major NFC pattern that has been reported in SLE patients was non-specific sub-types, followed by normal pattern and scleroderma pattern. In (SLE) patients are reported a large spectrum of antibodies, including the anti-ribonucleoproteins (RNP) antibodies These antibodies were linked to several clinical manifestations and prognostic in patients with SLE. Anti-U1-RNP antibodies are involved in both innate and adaptive immune responses during pathogenesis of connective tissue diseases 12. U1-RNP complex is an intra nuclear protein that converts pre-mRNA to mature RNA and constitutes three specific proteins A, C, and 70 kDa. High titer RNP antibodies are detected in MCTD patients and correlated with Clinical disease activity index and the frequent complication of pulmonary artery hypertension in those patients . It also has been found that NFC may detect subclinical microvascular changes in SLE in the presence of anti-U1-RNP antibodies and may facilitate early preventive therapy for major organ vasculopathy .

ELIGIBILITY:
Inclusion Criteria:

* Adult SLE Patients who fulfilled the 2012 systemic lupus international collaborating clinics (SLICC) criteria

Exclusion Criteria:

1. SLE patient aged less than 18 yeares old.
2. Individuals with other autoimmune diseases (rheumatoid arthritis dermatomyositis, scleroderma, mixed connective tissue disease).
3. Congestive cardic failure and presence of clupping.
4. Coexisting diabetes mellitus.
5. history of smoking.
6. Patients unable to co-operate for nailfold capillaroscopic examination

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: : Collected from Rheumatology, Rehabilitation and Physical Medicine Department, inpatient and outpatient clinics , Assiut University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Frequency of nail fold capillary changes in SLE patient. | baseline
  capillary changes on nailfold capillaroscopy examination for SLE patients

SECONDARY OUTCOMES:
1- Detection of patterns of nailfold capillary changes in SLE . | baseline
  to detect different patterns by nailfold capillaroscopy
2-Correlation of nailfold capillary changes in SLE patient and Anti-U1RNP antibodies. | baseline
  relation of Anti U1 RNP antibodies and microvasculature as detected by NFC examination
3-Correlation of nailfold capillary changes with SLE disease activity . | baseline
  relation of SLE disease activity and microvasculature as detected in NFC examination

REFERENCES:
- [Background] Zhao T, Lin FA, Chen HP. Pattern of Nailfold Capillaroscopy in Patients With Systemic Lupus Erythematosus. Arch Rheumatol. 2020 Apr 20;35(4):568-574. doi: 10.46497/ArchRheumatol.2020.7763. eCollection 2020 Dec. PMID 33758813
- [Background] Chebbi PP, Goel R, Ramya J, Gowri M, Herrick A, Danda D. Nailfold capillaroscopy changes associated with anti-RNP antibodies in systemic lupus erythematosus. Rheumatol Int. 2022 Aug;42(8):1355-1361. doi: 10.1007/s00296-021-04894-4. Epub 2021 Jun 2. PMID 34076720